CLINICAL TRIAL: NCT00168961
Title: Enteral Nutrition in Liver Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EE1
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2005-09

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis Child B or C
MeSH Terms: conditions — Liver Cirrhosis

INTERVENTIONS:
Dietary Supplement: High Protein Energy, Fresenius-Kabi (nutritional intervention)

SUMMARY:
Malnutrition is frequently occurring in patients with liver cirrhosis and is associated with a poorer outcome, as it determines life quality and affects both morbidity and mortality.

Long term prognosis after liver transplantation also depends on the nutritional status.

Therefore, the early diagnosis and intervention for malnutrition is an important issue in the clinical management of liver cirrhosis. However, oral intake has been shown to be insufficient due to disease related anorexia or concomitant drowsiness and confusion.

Specific aims: To investigate the effect of early nutritional intervention via tube feeding on nutritional status, functional status (hand grip strength and peak flow), life quality and disease related complications such as intestinal permeability, and oxidative stress, as well as liver function.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis (Child B or Child C)

Exclusion Criteria:

* Malignant comorbidity
* Encephalopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pirlich, MD, Principal Investigator — Charite Universitätsmedizin CCM Klinik für Gastroenterologie
Locations (1):
- Charite Universitätsmedizin Klinik für Gastroenterologie, Berlin, Germany